CLINICAL TRIAL: NCT04940026
Title: A Phase 1, Open-label, Single Center, One Period, One Sequence Study to Determine Absorption, Metabolism, and Excretion of a Single Oral Dose of Radiolabeled [14C]- SAR439859 and an Assessment of the Absolute Oral Bioavailability Using the Microdosing Technique in Healthy Post-menopausal Women
Brief Title: Study to Determine Absorption, Metabolism, and Excretion of [14C]-SAR439859, and to Assess Absolute Oral Bioavailability of Amcenestrant (SAR439859), in Healthy Post-menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BEX15859
Record Dates: First submitted 2021-06-14; First posted 2021-06-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Healthy Volunteers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAR439859 (Experimental): Single oral dose of SAR439859 at Day 1 in fasted condition followed by intravenous administration of [14C]-SAR439859 microtracer 3 hours later, and single oral dose of [14C]-SAR439859 at Day 7 in fasted condition
  Interventions: Drug: amcenestrant; Drug: [14C]-SAR439859 microtracer; Drug: [14C]-SAR439859

INTERVENTIONS:
Drug: amcenestrant — Tablet Oral
  Other Names: SAR439859
Drug: [14C]-SAR439859 microtracer — Solution for infusion Intravenous
Drug: [14C]-SAR439859 — Powder for oral solution Oral

SUMMARY:
Primary Objectives:

* To assess the excretion balance after oral and IV administration of [14C]-SAR439859
* To assess PK of total radioactivity, [14C] -SAR439859 and its metabolite (M7) after IV administration of [14C]-SAR439859 and, PK of radioactivity, SAR439859 and M7 after oral administration of SAR439859 alone or with [14C]-SAR439859
* To assess IV clearance and absolute bioavailability of SAR439859 using microdose of [14C]-SAR439859 tracer on top of a single tablet oral dose.
* To assess relative bioavailability of SAR439859 given as tablet or solution

Secondary objectives:

* To collect samples in order to assess metabolic profile in plasma and excreta of SAR439859 after oral administration of [14C]-SAR439859 as solution, contribution in plasma of SAR439859 and metabolite relative to total radioactivity and identify metabolites (samples will be analyzed according to metabolic analysis plan and results will be documented in a separate report).
* To assess safety and tolerance of SAR439859

DETAILED DESCRIPTION:
Total study duration is 3 to 10 weeks, including a screening period of up to 27 days, treatment period of up to 16 days and a follow-up and end of study of up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

Female participants (age between 40 and 75 years old) who are postmenopausal or had post-bilateral surgical oophorectomy not linked to a history of cancer.

Participants who are overtly healthy. Body weight within 40.0 and 95.0 kg and body mass index (BMI) within the range 18.0 and 30 kg/m2 (inclusive).

Capable of giving signed informed consent.

Exclusion Criteria:

Subject has clinical signs and symptoms consistent with COVID-19, e.g., fever, dry cough, dyspnea, loss of taste and smell, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening.

Subject who had severe course of COVID-19 (i.e., hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).

Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).

Blood donation, any volume (usually approximately 500 mL), within 2 months before inclusion.

Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.

History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day).

Smoking regularly more than 5 cigarettes or equivalent per week, unable to stop smoking during the study (occasional smoker can be enrolled).

Excessive consumption of beverages containing xanthine bases (more than 5 cups or glasses per day).

Subjects who are occupationally exposed to radiation as defined in the Ionizing Radiation Regulations 2017.

Participation in a trial with [13C] or [14C] radiolabeled medication in the 12 months preceding the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose, SAR439859 and M7 excreted in urine and feces after IV administration | Day 1 to Day 6
Percentage of radioactive dose excreted in urine and feces after oral administration | Day 7 up to max Day 44
Assessment of Pharmacokinetic (PK) parameter: AUC for radioactivity and SAR439859 after IV administration | Day 1 to Day 3
  Area under the plasma concentration versus time curve extrapolated to infinity
Assessment of PK parameter: t1/2z for radioactivity and SAR439859 after IV administration | Day 1 to Day 3
  Terminal half-life associated with the terminal slope (λz)
Assessment of PK parameter: CL for SAR439859 after IV administration | Day 1 to Day 3
  Total body clearance
Assessment of PK parameter: AUC ratios after IV administration | Day 1 to Day 3
  SAR439859 to radioactivity ratio for plasma AUC
Assessment of PK parameter: Cmax for radioactivity and SAR439859 after oral administration | Day 1 to Day 5, Day 7 to Day 11
  Maximum plasm concentration observed
Assessment of PK parameter: tmax for radioactivity and SAR439859 after oral administration | Day 1 to Day 5, Day 7 to Day 11
  Time to reach Cmax
Assessment of PK parameter: AUC for radioactivity and SAR439859 after oral administration | Day 1 to Day 5, Day 7 to Day 11
Assessment of PK parameter: t1/2z for radioactivity and SAR439859 after oral administration | Day 1 to Day 5, Day 7 to Day 11
Assessment of PK parameter: AUC ratios after oral administration | Day 7 to Day 11
  SAR439859 to radioactivity ratio for plasma AUC
Assessment of PK parameter: Cmax for M7 after IV and oral administration | Day 1 to Day 5, Day 7 to Day 11
Assessment of PK parameter: AUC for M7 after IV and oral administration | Day 1 to Day 5, Day 7 to Day 11
Assessment of PK parameter: t1/2z for M7 after IV and oral administration | Day 1 to Day 5, Day 7 to Day 11
Assessment of PK parameter: Rmet Cmax after IV and oral administration | Day 1 to Day 5, Day 7 to Day 11
  M7 to SAR439859 ratio for plasma Cmax
Assessment of PK parameter: Rmet AUC after IV and oral administration | Day 1 to Day 5, Day 7 to Day 11
  M7 to SAR439859 ratio for plasma AUC
Absolute oral bioavailability of SAR439859 | Day 1 to Day 5, Day 7 to Day 11
  Absolute oral bioavailability, expressed as a percentage, estimated from AUCs obtained after oral and IV administration
Relative bioavailability of SAR439859 after oral administration | Day 1 to Day 5, Day 7 to Day 11

SECONDARY OUTCOMES:
Number of participants with adverse events | Day 1 to Day 44

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site Number 8260001, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BEX15859 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25221&tenant=MT_SNY_9011